CLINICAL TRIAL: NCT03725709
Title: Metabolomic Profiling of Cerebrospinal Fluid and Plasma in Patients With type2 Diabetes
Brief Title: Metabolomic Profiling of in Patients With type2 Diabetes
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 140-9207A
Record Dates: First submitted 2018-09-27; First posted 2018-10-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2018-09

CONDITIONS: Diagnoses Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be centrifuged for 10 min at 4 °C and 4000 rpm. The supernatant (plasma) samples will be stored in aliquots at -80 °C until analysis. CSF samples will be stored in aliquots at -80 °C before analysis. The sample will be analyzed using hydrogen-1 nuclear magnetic resonance (1H-NMR) and lipid chromatography-mass spectrometry (LC-MS) in the Metabolomic Core Laboratory at Chang Gung Memorial Hospital or Chang Gung University. Demographic data including age, gender, body weight, blood pressure and past medical data will be investigated. Blood HbA1c, blood/CSF glucose and insulin level also will be measured.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: spinal anesthesia
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Plan to enroll 120 Type 2 diabetes and 120 non-diabetes patients with received spinal anesthesia.Blood will be collected at time point of pre-anesthesia 10 minutes and CSF samples will be collected at time point during spinal anesthesia induction. Blood will be collected, drawn into EDTA-coated tube.

SUMMARY:
To exam the metabolomic profiling of CSF and plasma in diabetes and establish the human CSF Metabolome Database of Type 2 DM.

DETAILED DESCRIPTION:
Human cerebral spinal fluid (CSF) is known to be a rich source of small molecule biomarkers for central neurological and neurodegenerative diseases. However, the metaboloic bases of CSF in diabetes patient have not been studied. In this plan, the investigators will use analytical platforms, including nuclear magnetic resonance (NMR), liquid chromatography-mass spectrometry (LC-MS), to perform quantitative metabolomics on human CSF and blood samples and further establish the human CSF Metabolome Database of DM. This work will can supply important CSF metabolic profit information and help to facilitate a wide range of metabolomic studies on central nervous system diseases and their associations disease.

ELIGIBILITY:
Inclusion Criteria:

Diabetes group

1. .20-75 years of age
2. .Type 2 diabetes patient by clinical diagnosis
3. .American Association of Anesthesiologists (ASA)≦III

Control group (non-diabetic group):

1. .20-75 years of age
2. .No history of DM and other systemic illness
3. .American Association of Anesthesiologists (ASA)≦ II

Exclusion Criteria:

1. patient refuses to sign informed consent
2. patients with coagulopathy, systemic infective disease and severe liver and renal function impairment.
3. patients with spine or brain tumor and severe CNS disease.
4. the presence of severe and/or uncontrolled and/or unstable medical disease within 12 months prior to study other than DM which could compromise participation in the study (e.g. acute pancreatitis, stroke, liver cirrhosis, congestive heart failure, and systemic immune disorder etc.
5. Concurrent participation or planning to participate in another interventional clinical trial (Concurrent participation in an observational trial allowed)

   -

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with received spinal anesthesia and had written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Find the reliable biomarkers, using metabolomic analysis [NMR, LC-MS] | Through study completion, an average of 1 year
  Use metabolomic analysis to connect CSF and blood metabolomic profiles information for further clarification of the influence of DM in CNS and expect to find new reliable biomarkers in diabetes patient for early predict DM progression and outcome.
Exam metabolic profiles of CSF and plasma in diabetes. (Metabolites analysis of CSF and plasma) | Through study completion, an average of 1 year
  Metabolites analysis of CSF and plasma will be investigated by NMR, LC-MS. Peak lists of all NMR and LC/MS/MS spectra will be searched against the database through a web server for metabolomic data analysis and further establish the CSF Metabolome Database.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan